CLINICAL TRIAL: NCT01788787
Title: Implementation of an Automated EMR System to Connect Smokers in a Safety Net Healthcare System With Smoking Cessation Treatment
Brief Title: Ask Advise Connect (AAC) Harris Heath CPRIT
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cancer Therapy and Research Center, Texas (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-1112; PP12019 (Other: Cancer Prevention and Research Institute of Texas (CPRIT))
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Tobacco Use Cessation
Keywords: Cancer Prevention; Tobacco Use Cessation; Ask Advise Connect; AAC; Smoking Cessation Treatment; Texas Quitline; Saliva sample; Telephone Counseling; Nicotine replacement; Interviews
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva sample to test for cotinine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Texas Quitline: Patients interested in smoking cessation treatment by calling the Texas Quitline.
  Interventions: Behavioral: Quitline-Delivered Proactive Telephone Counseling; Behavioral: Follow-Up Phone Call
- Training Providers: Medical staff (i.e., medical assistants, licensed vocational nurses, registered nurse and physicians).
  Interventions: Behavioral: Smoking Cessation Training; Behavioral: Qualitative Interviews Concerning the Implementation of AAC

INTERVENTIONS:
Behavioral: Quitline-Delivered Proactive Telephone Counseling — Smokers who enroll in treatment receive standard counseling protocol offered by the Quitline. This includes up to five proactive telephone counseling calls, each designed to provide practical expert support to help smokers develop problem-solving and coping skills, secure social support, and design a plan for successful cessation and long-term abstinence.
  Groups: Texas Quitline
Behavioral: Follow-Up Phone Call — Six months after enrolling in treatment with the Texas Quitline, an MD Anderson research team member will contact patients to assess their smoking status via telephone.
  Groups: Texas Quitline
Behavioral: Smoking Cessation Training — Medical staff (i.e., medical assistants, licensed vocational nurses, registered nurse and physicians) receive initial face-to-face group training on how to ask patients about their smoking status, advise them to quit, and connect them with the Quitline. The specific content of the session will include information on quitting smoking, how to implement AAC, the effectiveness of telephone counseling for smoking cessation delivered via quitlines, and pharmacotherapies including nicotine replacement.
  Groups: Training Providers
Behavioral: Qualitative Interviews Concerning the Implementation of AAC — MD Anderson staff conduct individual in-depth interviews with administrative leadership as well as those medical staff who are authorized to enter patient information into the EMR and are trained in the Ask-Advise-Connect approach. All in-depth interviews will be recorded and transcribed.
  Groups: Training Providers

SUMMARY:
The goal of this behavioral research study is to learn about the outcomes of smoking cessation treatment. Researchers want to learn how many smokers stopped smoking after taking part in smoking cessation treatment with the Texas Quitline.

DETAILED DESCRIPTION:
Study Test:

If you agree to take part in this study, you will collect a saliva sample to test for cotinine to confirm your smoking status. Cotinine is a chemical released in your body when it breaks down nicotine. You will receive a kit in the mail with supplies for the testing. The study staff will call you to make sure that you received the kit and to discuss the instructions with you. To collect the saliva, you will put a small piece of cotton in your mouth for a few minutes. You will mail the saliva sample back to the study staff, using a postage-paid envelope.

Length of Study:

Your participation in this study will be complete after you collect the saliva sample and mail it back to the study staff. Study data will be destroyed 5 years after the study has been completed and the data has been analyzed. Data collected in this study will not be used for future research.

This is an investigational study.

Up to 1,459 participants will be enrolled in this study. All will be enrolled at Harris Health System clinics.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Self-reported current smoker
3. Present for care at one of the 13 Harris Health System (HHS) community clinics
4. Has a working telephone number

Exclusion Criteria:

1) None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from the Harris Health System Community Health Clinics
Sampling Method: Non-Probability Sample
Enrollment: 5212 (Estimated)
Dates: Start 2013-04 (Actual); Primary Completion 2049-04 (Estimated); Study Completion 2049-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Reach of Ask Advise Connect (AAC) Smoking Cessation Program | 2 years
  Reach defined as the proportion of smokers that enroll in treatment with the Quitline. To evaluate the reach of AAC, we will calculate the proportion of smokers seen at the 13 Harris Health System community health clinics during the two-year treatment dissemination period that enroll in treatment with the Quitline.

SECONDARY OUTCOMES:
Efficacy of Ask Advise Connect (AAC) Smoking Cessation Program | 6 months
  Efficacy is defined as the proportion of smokers who agree to be connected to the Quitline that enroll in treatment who successfully achieve abstinence assessed 6 months following treatment enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna H. McNeill, PHD, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Harris Health System, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org